CLINICAL TRIAL: NCT03778177
Title: Mapping Towards a Cure - Identification of Neurophysiologic Signatures of Trigeminal Neuralgia Pain
Brief Title: Neurophysiologic Signatures of Trigeminal Neuralgia Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Facial Pain Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNP001
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Trigeminal Neuralgia (TN)
Keywords: transcranial electrical stimulation (tES)
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — TES

STUDY DESIGN:
Intervention Model Description: The investigators will use of transcranial electrical stimulation (tES) to evaluate pain in patients with Trigeminal Neuralgia (TN).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trigeminal Neuralgia Pain Diagnosis (Experimental): Healthy patients between the ages of 18-75 who have been diagnosed with moderate to severe Trigeminal Neuralgia Pain. The study team will perform transcranial electrical brain stimulation using either electrodes that are in the form of two salt-water soaked sponges attached to the head or a set of smaller gel-covered disk electrodes that fit inside the electrode holders of the EEG cap. During stimulation a weak direct or alternating current will be passed through the stimulating electrodes. Stimulation may last 20 to 30 minutes.
  Interventions: Procedure: transcranial electrical brain stimulation

INTERVENTIONS:
Procedure: transcranial electrical brain stimulation — Pain ratings will be recorded before and after transcranial brain electrical stimulation procedures using a Visual Analog Scale (VAS).
  Other Names: tES

SUMMARY:
Trigeminal neuralgia (TN) is an idiopathic pain disorder that is characterized by episodic attacks of intense facial pain, described as paroxysms of stabbing, electric, or explosive pain, and lasting for a few seconds or longer, often producing a tic-like facial movement, and can occur up to hundreds of times per day. This pain is known to be one of the worst pain conditions that a patient can suffer and has been called the "suicide disease". Given the severity of this disorder, determining the cause becomes essential for finding a cure. This project will study the cause of TN using a translational approach, which means the research project will be completed in both humans and animals. The investigators hypothesize that there are specific areas of the brain and spinal cord that will provide a "signature" center of activity. The study team will use state of the art magnetic resonance imaging (MRI) machines and other non-invasive brain activity measurements, including electroencephalography (EEG) to locate these centers in people with TN before and after their pain has started. Recent studies have investigated the effects of transcranial electrical stimulation (tES) for pain control. Transcranial electrical stimulation (tES) includes transcranial direct current stimulation (tDCS) and transcranial alternating current stimulation (tACS). This approach is important because identifying similar regions neural activity will allow for us to study novel therapies in search of the cure for TN and this study has thus both basic and clinical neuroscience significance.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is an extremely painful and highly disabling orofacial pain disorder, often referred to as the "suicide disease," for which presently available therapies are largely ineffective or inadequate. Both the unpredictable response to treatment and variability in long-term clinical outcomes in TN strongly suggest that a range of peripheral and central mechanisms remain to be understood. The long-term goal is to identify the mechanisms involved in the initiation and progression of TN, and uncover rational targets for the safe and effective treatment of TN. The objective of this application is to explore the use of multimodal neuroimaging and neurophysiologic techniques in defining neural signatures of the disease. Additionally, the study team wants to evaluate the efficacy of transcranial electrical stimulation on relieving pain. The rationale for the proposed research is that identification of signature peripheral and central activation sites will allow for individualized treatment strategies for TN patients.

To modulate brain activities the investigators will use transcranial electrical stimulation (tES). tES is an emerging neuromodulation technique that can be noninvasively and safely applied in humans. tES can help better understand the causal roles of brain networks and brain activities and has shown efficacy in improving pain. tES has two main variations: transcranial direct current stimulation (tDCS) and transcranial alternating current stimulation (tACS). The former applies a weak direct current to the scalp whereas the latter applies a weak sinusoidal current to the scalp. tDCS can modulate the excitability of tissues under the stimulating electrodes. tACS is particularly suited for interacting with various oscillatory activities in the brain. tES has been used to study normal brain function and treat neurological and pain disorders as well. There is demonstrated efficacy in improvement of pain in subjects suffering from fibromyalgia and neuropathic pain. The study team will use different tDCS/tACS montages targeting different brain regions and observe behavior and neuronal activities. The current strength will be within 1mA or 2mA which has been shown to be safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who have been diagnosed with trigeminal neuralgia (TN) pain (ASA status 1, 2, or 3).
* Subjects diagnosed with TN pain must have average pain in the moderate to severe (Visual Analog Scale (VAS) of 30-100 mm) range. These subjects will be asked to stop their current medications for 24 hours prior to their scan.
* Patients diagnosed with classical trigeminal neuralgia, type 1 [TN1, G50.00], or symptomatic trigeminal neuralgia [TN2, G53.80] according to the International Classification of Headache (IHS) Disorders criteria (7).

Exclusion Criteria:

* Patients diagnosed with post-herpetic neuralgia, trigeminal neuropathic pain, and trigeminal deafferentation pain.
* TN subjects with ASA status 4-5 and Emergency operation.
* Presence of chronic disease (e.g. cardiovascular disease, liver disease, kidney disease, diabetes, etc.), other than trigeminal neuralgia.
* Pregnant females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Effects of transcranial electrical stimulating (tES) on pain. | Day 1
  Pain will be measured by subjects using a visual analog scale (VAS). The VAS is a psychometric measuring instrument presented as a 100-mm horizontal line anchored on one end with the words "no pain at all" which is 0 and at the other end with the words "worst pain imaginable" which is 100. Subjects will be asked to rate their pain on the VAS from 0-100 once before the stimulation and again after the stimulation is complete. The two scores will be compared to see if there is any reduction in subject's pain after the stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: John K Neubert, DDS, MS, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health Shands Hospital, Gainesville, Florida
  - McKnight Brain Institute, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad S, Galetta S. Trigeminal neuralgia: historical notes and current concepts. Neurologist. 2009 Mar;15(2):87-94. doi: 10.1097/NRL.0b013e3181775ac3. PMID 19276786
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Apr 13;4(4):CD008208. doi: 10.1002/14651858.CD008208.pub5. PMID 29652088
- [Background] Chaieb L, Antal A, Pisoni A, Saiote C, Opitz A, Ambrus GG, Focke N, Paulus W. Safety of 5 kHz tACS. Brain Stimul. 2014 Jan-Feb;7(1):92-6. doi: 10.1016/j.brs.2013.08.004. Epub 2013 Sep 13. PMID 24064065
- [Background] Saltychev M, Laimi K. Effectiveness of repetitive transcranial magnetic stimulation in patients with fibromyalgia: a meta-analysis. Int J Rehabil Res. 2017 Mar;40(1):11-18. doi: 10.1097/MRR.0000000000000207. PMID 27977465
- [Background] Lefaucheur JP. The use of repetitive transcranial magnetic stimulation (rTMS) in chronic neuropathic pain. Neurophysiol Clin. 2006 May-Jun;36(3):117-24. doi: 10.1016/j.neucli.2006.08.002. Epub 2006 Aug 23. PMID 17046606
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276